CLINICAL TRIAL: NCT02678663
Title: Randomized Comparison of Injection-Assisted Cold Snare Polypectomy Versus Endoscopic Mucosal Resection for Small (6-10mm) Colorectal Polyps
Brief Title: Injection-Assisted Cold Snare Polypectomy Versus Endoscopic Mucosal Resection for Small Colorectal Polyps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benizelion General Hospital (Other)
Responsible Party: Principal Investigator, Gregorios A. Paspatis, Director, Benizelion General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1513/3.2.2016
Record Dates: First submitted 2016-02-03; First posted 2016-02-10 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Colonic Polyps
Keywords: Colon polyp; Polypectomy; Cold snare; Endoscopic mucosal resection
MeSH Terms: conditions — Colonic Polyps | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Injection-assisted cold snare polypectomy (I-CSP) (Experimental): Polyps in this group will be resected with the cold snare technique after pre-lift of the lesion with a submucosal injection of methylene blue-tinted normal saline solution. The polyp and a small rim of normal tissue will be then snared closely and removed in a single piece without the use of electrocautery.
  Interventions: Procedure: Injection-assisted Cold Snare Polypectomy
- Endoscopic mucosal resection (EMR). (Active Comparator): Polyps in this group will be removed in a single piece by using an "inject-and-cut" EMR technique. Methylene blue-tinted normal saline solution will be injected into the submucosal space followed by the application of snare cautery for lesion resection.
  Interventions: Procedure: Endoscopic Mucosal Resection

INTERVENTIONS:
Procedure: Injection-assisted Cold Snare Polypectomy — Resection of a polyp after blue-tinted saline injection using a cold snare (without application of electrocautery)
  Arms: Injection-assisted cold snare polypectomy (I-CSP)
Procedure: Endoscopic Mucosal Resection — Resection of a polyp after blue-tinted saline injection using snare electrocautery
  Arms: Endoscopic mucosal resection (EMR).

SUMMARY:
Complete resection of neoplastic polyps is pivotal, as 8.8% to 50% of interval cancers may arise as a consequence of incomplete polypectomy. However, the ideal method to remove small colorectal polyps remains uncertain. The investigators designed a randomized controlled trial to assess whether injection-assisted cold snare polypectomy may be noninferior to EMR for the resection of small (6-10mm) colorectal polyps.

DETAILED DESCRIPTION:
Polypectomy is the basis of colorectal cancer prevention by interrupting the adenoma-to-carcinoma sequence. Most of the polypectomies are performed for diminutive (≤5mm) or small (6-10mm) colorectal lesions which represent >90% of the overall burden of resected polyps. Although the potential for neoplasia is usually size-dependent, recent evidence suggested that even diminutive and small polyps harbor a substantial risk of advanced neoplasia (in some series as high as 9-10%). Complete resection of neoplastic polyps is pivotal, as 8.8% to 50% of interval cancers may arise as a consequence of incomplete polypectomy. However, the ideal method to remove small colorectal polyps remains uncertain. Cold snare polypectomy has become standard technique allowing for comprehensive and safe resection of diminutive polyps, though significant incomplete resection rates have challenged the implementation of CSP for larger (in particular 8-10mm) polyps. Submucosal injection of a solution containing a staining dye could improve the outcome of cold snare polypectomy: a) lift of the lesion with submucosal chromoendoscopy could sharply delineate margins and facilitate capture and removal by using a cold snare, and b) formation of a submucosal cushion could minimize mechanical damage to the submucosal vessels, preventing the occurrence of immediate bleeding.

Use of electrocautery is believed to reduce the risk of incomplete resection, although it is less attractive from a safety standpoint due to the risk of complications including delayed bleeding, post-polypectomy syndrome and perforation. Injection of a submucosal solution in order to lift the lesion (injection-assisted endoscopic mucosal resection, EMR) facilitates "hot" resection of sessile or flat neoplasms and allows for a deeper resection margin as compared to conventional polypectomy, while it minimizes electrocautery damage by creating a safety cushion. Despite it is highly efficient, EMR still carries a substantial risk of complications (in most series 7-8%) which has generally limited uptake of the technique among endoscopists for the removal of small polyps.

Therefore, the investigators designed a randomized controlled trial to assess whether injection-assisted cold snare polypectomy may be noninferior to EMR for the resection of small (6-10mm) colorectal polyps.

METHODS

The study will be conducted in the endoscopy units of the Benizelion General Hospital (Heraklion, Crete, Greece) and the Konstantopoulio General Hospital (Nea Ionia, Athens, Greece). Consecutive subjects over the age of 18 years who agree informed consent and who have at least one polyp of eligible size (6-10mm) will be randomly assigned in two groups:

1. Injection-assisted cold snare polypectomy (I-CSP). Polyps in this group will be resected with the cold snare technique after pre-lift of the lesion with a submucosal injection of methylene blue-tinted normal saline solution. The polyp and a small rim of normal tissue will be then snared closely and removed in a single piece without the use of electrocautery.
2. Endoscopic mucosal resection (EMR). Polyps in this group will be removed in a single piece by using an "inject-and-cut" EMR technique. Methylene blue-tinted normal saline solution will be injected into the submucosal space followed by the application of snare cautery for lesion resection.

All polypectomy specimens will be retrieved by suctioning into a polyp trap or by using retrieval forceps and send for histopathological examination.

The polypectomy site will be rinsed with tap water and carefully inspected for residual polyp. Targeted biopsies will be obtained from any areas in the polypectomy site margin suspicious for residual tissue. Protrusions in the polypectomy base after I-CSP will be recorded and a biopsy will be taken for separate histological assessment.

Histological evaluation of polypectomy specimens and post-polypectomy biopsy specimens will rely on the criteria of the World Health Organization and will be performed by experienced GI pathologists blinded to the polytectomy technique used and the endoscopic findings.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over the age of 18 years who agree informed consent and who have at least one polyp of eligible size (6-10mm)

Exclusion Criteria:

* Anticoagulant therapy during the past 1 week of the procedure
* Known coagulopathy
* History of liver cirrhosis, chronic kidney disease, malignancy, inflammatory bowel disease, significant infectious disease, polyposis syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2016-01; Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Complete Resection Rate | Two weeks after each polypectomy

SECONDARY OUTCOMES:
Incidence of complications (intraprocedural bleeding, postprocedural bleeding, post-polypectomy syndrome, perforation). | Two weeks after each polypectomy
Necessity of hemostasis (due to intraprocedural or postprocedural bleeding) | Two weeks after each polypectomy
Polyp retrieval rate | Two weeks after each polypectomy

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Konstantopoulio General Hospital, Nea Ionia, Athens
  - Benizelion General Hospital, Heraklion, Crete

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Papastergiou V, Paraskeva KD, Fragaki M, Dimas I, Vardas E, Theodoropoulou A, Mathou N, Giannakopoulos A, Karmiris K, Mpitouli A, Apessou D, Giannikaki L, Karagiannis JA, Chlouverakis G, Paspatis GA. Cold versus hot endoscopic mucosal resection for nonpedunculated colorectal polyps sized 6-10 mm: a randomized trial. Endoscopy. 2018 Apr;50(4):403-411. doi: 10.1055/s-0043-118594. Epub 2017 Sep 12. PMID 28898922